CLINICAL TRIAL: NCT00051350
Title: Macronutrients and Cardiovascular Risk
Brief Title: OmniHeart Trial: Macronutrients and Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00069360; R01HL067098 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-13 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Hypertension | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Individuals were randomized to a sequence of 3 diets (CARB, UNSAT, PROTEIN)
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were unaware of diet sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CARB (Placebo Comparator): Diet rich in carbohydrate
  Interventions: Other: CARB
- UNSAT (Active Comparator): Diet rich in unsaturated fat
  Interventions: Other: CARB
- PROTEIN (Active Comparator): Diet rich in protein
  Interventions: Other: CARB

INTERVENTIONS:
Other: CARB
  Other Names: UNSAT; PROTEIN

SUMMARY:
To compare the effects on blood pressure and plasma lipids of three different diets--a carbohydrate-rich diet, a protein-rich diet, or a diet rich in unsaturated fat.

DETAILED DESCRIPTION:
BACKGROUND:

While there is widespread consensus that the optimal diet to reduce cardiovascular risk should be low in saturated fat, the type of macronutrient that should replace saturated fat (carbohydrate, protein or unsaturated fat) is a major, unresolved research question with substantial public health implications. The study will evaluate these three dietary approaches by studying their effects on established coronary risk factors and a selected group of emerging risk factors.

DESIGN NARRATIVE:

The study design was a randomized, three period cross-over feeding study that compared the effects on blood pressure and plasma lipids of a carbohydrate-rich diet patterned after the DASH diet (CARB) to two other diets, one rich in protein (PROTEIN) and another rich in unsaturated (UNSAT) fat, predominantly monounsaturated fat. The DASH diet has been shown to reduce blood pressure and LDL-cholesterol substantially, and is currently recommended by policy makers. During a one week run-in, all participants were fed samples of the three study diets (CARB, PROTEIN and UNSAT). Using a three period cross-over design, participants were then randomly assigned to the CARB, PROTEIN or UNSAT diet. Each feeding period lasted six weeks; a washout period of at least two weeks separated each feeding period. Throughout feeding (run-in and the three intervention periods), participants were fed sufficient calories to maintain their weight. Trial participants were 30 years of age or older, with systolic blood pressure of 120-159 mmHg or diastolic blood pressure of 90-99 mmHg. Primary outcomes variables were blood pressure and the established plasma lipid risk factors (LDL-C, HDL-C and triglycerides). Secondary outcomes include total cholesterol, apolipoproteins VLDL-apoB, VLDL-apoCIII, apolipoprotein B, non-HDL cholesterol, and lipoprotein(a).

ELIGIBILITY:
Inclusion criteria:

* Healthy adults
* Aged 30 years and older
* Systolic blood pressure of 120 to 159 mm Hg or a diastolic blood pressure of 80 to 99 mm Hg.

Exclusion criteria:

* Diabetes
* Active or prior Cardiovascular disease (CVD)
* LDL cholesterol greater than 220 mg/dL (>5.70 mmol/L)
* Fasting triglycerides greater than 750 mg/dL (>8.48 mmol/L)
* Weight more than 350 lb (>159 kg)
* Taking medications that affect blood pressure or blood lipid levels
* Unwillingness to stop taking vitamin and mineral supplements
* Alcoholic beverage intake of more than 14 drinks per week.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Appel, Study Chair — Johns Hopkins University

REFERENCES:
- [Background] Appel LJ, Sacks FM, Carey VJ, Obarzanek E, Swain JF, Miller ER 3rd, Conlin PR, Erlinger TP, Rosner BA, Laranjo NM, Charleston J, McCarron P, Bishop LM; OmniHeart Collaborative Research Group. Effects of protein, monounsaturated fat, and carbohydrate intake on blood pressure and serum lipids: results of the OmniHeart randomized trial. JAMA. 2005 Nov 16;294(19):2455-64. doi: 10.1001/jama.294.19.2455. PMID 16287956
- [Derived] Zhang B, Furtado JD, Andraski AB, Guglielmo B, Appel LJ, Wang K, Yasunaga S, Saku K, Ikewaki K, Sacks FM. Partially Replacing Dietary Carbohydrate With Unsaturated Fat or Protein Shifts Protein-Based HDL Subspecies Toward Lower Coronary Heart Disease Risk. Arterioscler Thromb Vasc Biol. 2026 Jan;46(1):251-267. doi: 10.1161/ATVBAHA.125.323709. Epub 2025 Dec 2. PMID 41328959
- [Derived] Kim H, Lichtenstein AH, Ganz P, Miller ER 3rd, Coresh J, Appel LJ, Rebholz CM. Associations of circulating proteins with lipoprotein profiles: proteomic analyses from the OmniHeart randomized trial and the Atherosclerosis Risk in Communities (ARIC) Study. Clin Proteomics. 2023 Jul 3;20(1):27. doi: 10.1186/s12014-023-09416-x. PMID 37400771
- [Derived] Belanger MJ, Wee CC, Mukamal KJ, Miller ER, Sacks FM, Appel LJ, Shmerling RH, Choi HK, Juraschek SP. Effects of dietary macronutrients on serum urate: results from the OmniHeart trial. Am J Clin Nutr. 2021 Jun 1;113(6):1593-1599. doi: 10.1093/ajcn/nqaa424. PMID 33668058
- [Derived] Zhang M, Juraschek SP, Appel LJ, Pasricha PJ, Miller ER 3rd, Mueller NT. Effects of High-Fiber Diets and Macronutrient Substitution on Bloating: Findings From the OmniHeart Trial. Clin Transl Gastroenterol. 2020 Jan;11(1):e00122. doi: 10.14309/ctg.0000000000000122. PMID 31972610
- [Derived] Mueller NT, Zhang M, Juraschek SP, Miller ER, Appel LJ. Effects of high-fiber diets enriched with carbohydrate, protein, or unsaturated fat on circulating short chain fatty acids: results from the OmniHeart randomized trial. Am J Clin Nutr. 2020 Mar 1;111(3):545-554. doi: 10.1093/ajcn/nqz322. PMID 31927581
- [Derived] Kovell LC, Yeung EH, Miller ER 3rd, Appel LJ, Christenson RH, Rebuck H, Schulman SP, Juraschek SP. Healthy diet reduces markers of cardiac injury and inflammation regardless of macronutrients: Results from the OmniHeart trial. Int J Cardiol. 2020 Jan 15;299:282-288. doi: 10.1016/j.ijcard.2019.07.102. Epub 2019 Aug 2. PMID 31447226
- [Derived] Loo RL, Zou X, Appel LJ, Nicholson JK, Holmes E. Characterization of metabolic responses to healthy diets and association with blood pressure: application to the Optimal Macronutrient Intake Trial for Heart Health (OmniHeart), a randomized controlled study. Am J Clin Nutr. 2018 Mar 1;107(3):323-334. doi: 10.1093/ajcn/nqx072. PMID 29506183
- [Derived] Juraschek SP, Miller ER 3rd, Appel LJ, Christenson RH, Sacks FM, Selvin E. Effects of dietary carbohydrate on 1,5-anhydroglucitol in a population without diabetes: results from the OmniCarb trial. Diabet Med. 2017 Oct;34(10):1407-1413. doi: 10.1111/dme.13391. Epub 2017 Jul 9. PMID 28574153
- [Derived] Haring B, von Ballmoos MC, Appel LJ, Sacks FM. Healthy dietary interventions and lipoprotein (a) plasma levels: results from the Omni Heart Trial. PLoS One. 2014 Dec 15;9(12):e114859. doi: 10.1371/journal.pone.0114859. eCollection 2014. PMID 25506933
- [Derived] Gadgil MD, Appel LJ, Yeung E, Anderson CA, Sacks FM, Miller ER 3rd. The effects of carbohydrate, unsaturated fat, and protein intake on measures of insulin sensitivity: results from the OmniHeart trial. Diabetes Care. 2013 May;36(5):1132-7. doi: 10.2337/dc12-0869. Epub 2012 Dec 5. PMID 23223345
- [Derived] Juraschek SP, Appel LJ, Anderson CA, Miller ER 3rd. Effect of a high-protein diet on kidney function in healthy adults: results from the OmniHeart trial. Am J Kidney Dis. 2013 Apr;61(4):547-54. doi: 10.1053/j.ajkd.2012.10.017. Epub 2012 Dec 4. PMID 23219108
- [Derived] Furtado JD, Campos H, Sumner AE, Appel LJ, Carey VJ, Sacks FM. Dietary interventions that lower lipoproteins containing apolipoprotein C-III are more effective in whites than in blacks: results of the OmniHeart trial. Am J Clin Nutr. 2010 Oct;92(4):714-22. doi: 10.3945/ajcn.2009.28532. Epub 2010 Sep 8. PMID 20826623